CLINICAL TRIAL: NCT01604096
Title: Doctors and Local Media: a Synergy for Public Health Information? A Controlled Trial to Evaluate the Effects of a Multifaceted Campaign on Antibiotic Prescribing
Brief Title: Controlled Trial to Evaluate a Local Information Campaign on Antibiotic Prescribing in Italy
Acronym: LOCAAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Health and Social Care Agency, Italy (Other Government)
Collaborators: Local Health Authority, Parma (Unknown); Local Health Authority, Modena (Unknown); Change Institute, Turin (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: FARM8FKC3H
Record Dates: First submitted 2012-05-17; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Information; campaign; antibiotics; bacterial resistance; primary care
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention areas (Experimental): Provinces of Modena and Parma (about 1.100.000 inhabitants - campaign targeted to the general population), in Northern Italy (Emilia-Romagna Region)
  Interventions: Other: Multifaceted information campaign
- Control (No Intervention): All the other provinces in the Emilia-Romagna Region (where the information campaign has not been implemented)

INTERVENTIONS:
Other: Multifaceted information campaign — Following is the description of the multifaceted intervention:
  * brochures targeted at the general population and available in general practices, pharmacies, local health services and on the web (also translated in eight languages)
  * posters (same distribution as brochures)
  * short videos transmitted in local TVs, websites of Local Health Authorities and in video terminals in some pharmacies
  * radio-spots transmitted in local radio stations
  * advertisements in local newspapers
  * banners on websites of local newspapers
  * newsletter on antibiotic resistance in Emilia- Romagna, available to physicians and pharmacists
  * training courses in counselling strategies, directed to a subgroup of GPs and paediatricians
  Arms: Intervention areas

SUMMARY:
Use of information campaigns and educational interventions directed to citizens and supported by physicians, aimed at promoting the appropriate use of medicines, have been evaluated by several studies with conflicting results. These interventions are potentially relevant, favouring the reduction of unnecessary use of medicines and related risks. Several studies have specifically evaluated the promotion of the appropriate use of antibiotics in adults and children, with variable results. A controlled study has been proposed to evaluate the feasibility and effectiveness of a multifaceted intervention aimed at reducing antibiotic prescription by increasing awareness on risks of their unnecessary use.

Information has been provided to citizens through several media (posters, local TV, radio and newspapers, video terminals, websites of Local Health Authorities). Brochures with information on expected benefits and risks of antibiotics has also been available, either with direct access in waiting rooms and pharmacies or handed out and mediated by doctors. Physicians and pharmacists received specific data on local antibiotic resistance. A small group of representative doctors have also actively participated in defining the campaign key messages. A sample of general practitioners and paediatricians have been trained in patient counselling strategies.

The information campaign has been implemented in two Provinces of Emilia-Romagna during the fall-winter season (November 2011-February 2012). Change in the overall prescribing rate of antibiotics (expressed as DDD per 1000 inhabitants/day) in the intervention area will be compared versus other areas in the same Region. Knowledge and attitudes of the general population will be evaluated through a phone and internet survey on a representative sample.

This study could observe a reduction lower than 5% in the prescribing rate of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* the campaign has been targeted at the general population in the intervention areas

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Prescribing rate of antibiotics | up to 03/12
  Cumulative five-month changes in DDD per 1000 inhabitants/day of specific classes of antibiotics (J01C, J01D, J01F, J01M ATC codes) in general practice

SECONDARY OUTCOMES:
Antibiotic prescribing trends | up to 04/13
  Changes in antibiotic prescribing trends in eighteen months (same ATCs as for primary outcome)
Antibiotic expenditure | up to 03/12
  Changes in antibiotic expenditure per 1000 inhabitants/day (same ATCs as for primary outcome)
Knowledge/attitudes of the general population | up to 02/12
  Knowledge of and attitudes about the campaign messages, through a telephone and internet survey on a sample of the target population.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Formoso, MPH, MPharm, Principal Investigator — Regional Health and Social Care Agency, Emilia Romagna Region (Italy)
Locations (2):
- Italy (2):
  - Local Health Authority of Modena, Modena
  - Local Health Authority of Parma, Parma

REFERENCES:
- [Background] LOcal Campaign on Antibiotics ALliance (LOCAAL) study group. Doctors and local media: a synergy for public health information?: a controlled trial to evaluate the effects of a multifaceted campaign on antibiotic prescribing (protocol). BMC Public Health. 2011 Oct 19;11:816. doi: 10.1186/1471-2458-11-816. PMID 22011332
- [Derived] Formoso G, Paltrinieri B, Marata AM, Gagliotti C, Pan A, Moro ML, Capelli O, Magrini N; LOCAAL Study Group. Feasibility and effectiveness of a low cost campaign on antibiotic prescribing in Italy: community level, controlled, non-randomised trial. BMJ. 2013 Sep 12;347:f5391. doi: 10.1136/bmj.f5391. PMID 24030722
- See also: Published protocol — http://www.biomedcentral.com/1471-2458/11/816
- See also: Campaign home page — http://www.ceveas.it/flex/cm/pages/ServeBLOB.php/L/IT/IDPagina/354